CLINICAL TRIAL: NCT02997813
Title: Assessment of Mobilization Cost for Multiple Myeloma Using 2 Different Mobilization Strategies: High-dose Cyclophosphamide Versus Plerixafor
Brief Title: Assessment of Mobilization Cost for Multiple Myeloma Using 2 Different Mobilization Strategies
Acronym: MOZOBIL
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Other Study IDs: IFM2014-05
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma; Blood Stem Cell Transplant Failure
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: All consecutive patients with complete set of data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and plerixafor
- Cohort 2: All consecutive patients with complete data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and cyclophosphamide

SUMMARY:
This is a retrospective observational cohort database analysis. The study will review retrospectively the records of patients undergoing a first peripheral blood stem cell mobilization for multiple myeloma in the databases from approximately 15 hospitals which are part of the IFM collaborative group. Patient records will be divided into two groups of 50 patients minimum, maximum 100 patients or up to the number of patient records that could be extracted. The first group of patients will have received plerixafor plus G-CSF without the administration of chemotherapy as a mobilization strategy and a second group of patients will have received cyclophosphamide plus G-CSF as a mobilization strategy.

All consecutive patients with complete set of data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and plerixafor and all consecutive patients with complete data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and cyclophosphamide will be included.

All data that will be analyzed will be extracted from the selected IFM institutions which are located in France.

ELIGIBILITY:
Inclusion Criteria:

* Hematology patients diagnosed with Multiple Myeloma who are candidates for autologous hematopoietic stem cell transplantation (ASCT) upfront.
* Age > 18 years
* Undergone prior successful peripheral blood stem cell mobilization with Cyclophosphamid or Plerixafor

Exclusion Criteria:

* Age < 18 years;
* Primary diagnosis other than Multiple Myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first group of patients will have received plerixafor plus G-CSF without the administration of chemotherapy as a mobilization strategy and a second group of patients will have received cyclophosphamide plus G-CSF as a mobilization strategy.
  All consecutive patients with complete set of data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and plerixafor and all consecutive patients with complete data (and who underwent apheresis) treated between 2009 and 2013 with G-CSF and cyclophosphamide will be included.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total cost of stem cell mobilization procedure (including remobilisation if applicable) | 2009-2013

SECONDARY OUTCOMES:
Number of visits for administration of mobilizing agents | 2009-2013
Duration (days) of administration of mobilizing agents | 2009-2013
Agents used as mobilizing agents | 2009-2013
Attainment of CD34+ target (yes, no) (min 2.106 cells/kg, ideal >4.106cells/kg) | 2009-2013
Number of days needed to meet CD34+ target level (min 2.106 cells/kg, ideal >4.106cells/kg) | 2009-2013

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Leleu, Dr, Study Chair — Service des maladies du sang, Hôpital Huriez, CHRU, Lille; Denis Caillot, Dr, Study Director — Service d'Hématologie Clinique, Hôpital Le Bocage, CHU Dijon; Eric Deconinck, Pr, Study Director — Hématologie, Hôpital Jean Minjoz, CHU Besançon; Samuel Limat, Pr, Study Director — Pharmacie centrale, Hôpital Jean Minjoz, CHU Besançon
Locations (9):
- France (9):
  - CHRU Dijon, Dijon
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - CHRU Hôtel Dieu, Nantes
  - Institut Curie Centre de Lutte Contre le Cancer (CLCC), Paris
  - La Pitié Salpetriêre, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Robert Debré Hématologie, Reims
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No